

# Study Information and Consent to Participate at Time 1

# PLEASE SCROLL DOWN TO LEARN ABOUT THIS STUDY AND CONSENT TO PARTICIPATE. ONCE YOU SELECT THE CONSENT BUTTON YOU WILL BE TAKEN TO THE SURVEY.

#### What is this study about?

The Measurement-Based Transition Assistance (MBTA) Study will evaluate an online tool created for veterans who have transitioned from the military to civilian life within the past two years, though, we may offer this tool to all veterans in the future. The purpose of the online tool is to help veterans improve their well-being in different aspects of their lives as they transition from military to civilian life and to connect them with relevant supports. The tool focuses on four well-being related domains: vocation (i.e., employment, education, and caregiving), finances, health (i.e., physical and mental health), and social well-being.

#### Who are the collaborators on this study?

| This study is being funded and conducte | d by the VA. The online tool and study surveys are being hosted by |
|---|---|
| on behalf of VA. | is assisting with mailing of study invitations and reminders on |
| behalf of VA | |

## What does this study involve?

Over a period of approximately 3 months, participating veterans will complete two separate online surveys that will help us determine whether the online tool is helpful for veterans and for whom the online tool may be most helpful. The first survey will be completed today and the follow-up survey will be completed approximately 3 months from now. Each survey will take about 45 minutes to complete. Participants will be randomly assigned to try out the online tool either during the first timepoint (today) OR during a follow-up timepoint approximately three months later. Trying out the online tool includes completing a wellbeing assessment and receiving a report with feedback on your wellbeing as well as recommended resources for improving different aspects of your well-being.

### What kinds of questions are included in the study surveys?

You will be asked a series of questions about your background, personal traits, health, well-being, and well-being related behaviors and thoughts. We will also ask you for your thoughts about the online tool at the timepoint you receive it.

## Why do you want me to participate? How did you get my name?

Your name was obtained from VA records for the sole purpose of inviting you to participate in this research study. Your participation is completely voluntary. Our goal is to include men and women who have transitioned from military to civilian life within the past two years. We are seeking veterans with all types of military experiences and backgrounds — including veterans with different lengths of military service and racial/ethnic backgrounds. While we hope you will want to complete this survey as well as the 3-month follow-up survey, completing today's survey does not obligate you to complete the 3-month follow-up survey.

### Do I have to participate? Will participating or not affect the services or benefits I get from the VA?

No. Participation is completely up to you. If you decide not to participate, it will not affect your VA benefits or access to services in any way. By clicking the "I consent/agree to participate" button and completing this online survey, you are agreeing to participate in this study. If you choose not to participate, you may exit this webpage.

## Will my responses to study questions be kept private?

Yes. All information from study surveys and the online tool will be kept private. In order to help us keep your information private, we ask that you do not type your name or other identifying information (e.g., address) in response to study questions. Your responses will be combined with those of approximately 150 other recent veterans who

complete the same survey, and the survey results will be de-identified such that no individual can be identified. Your personally identifiable information will not be used in any reports.

| What steps are taken to ensure my privacy | aken to ensure my privacy? |
|-------------------------------------------|----------------------------|
|-------------------------------------------|----------------------------|

## Who has access to my information?

Your contact information was then given to participate in this research study. Your contact information was then given to participate in this research study, your contact information was then given to private the variety of the variety of participating in this study, your information will not be used for any other purposes. Only the company hosting the study surveys and online tool) and the study team at VA Boston Healthcare System will have access to your survey responses, which will be maintained separate from your names and other identifying information. Our study team has taken extensive measures to protect your privacy and ensure your confidentiality, as described previously. Please be assured that this information will not be shared with anyone else for any reason.

## What are the benefits and risks of participating in this study?

Participation in this study will help us learn from you and others whether our online tool may be beneficial to veterans transitioning out of the military. You will have the opportunity to try out the online tool, which may help you improve your well-being.

The risks associated with completing this study are minimal. There are two main risks. First, you may experience feelings of distress while responding to questions, such as questions that ask about your well-being. If some questions feel too personal or distressing, it is okay to skip them. If you would like to talk with someone about how this study makes you feel, please see the list of helpful phone numbers below. The other risk is a loss of privacy. However, as explained above, we have taken a number of steps to protect your privacy.

### Will I be compensated for participating in the survey?

If you complete this survey, you will receive a \$25 Amazon gift card. You will receive an additional \$25 Amazon gift card if you complete the 3-month follow-up survey. You can receive up to \$50 for completing both surveys.

## Who can I talk to if I still have questions?

If you have any questions about this project or your participation, please call the Principal Investigator of this study, Dr. at a large and If you call in the evenings or on weekends, feel free to leave a message. We will get back to you as soon as possible.

Other Helpful Phone Numbers (which you can call even if you don't take part in the study)

- If you feel distressed or you want to talk to someone about how you feel, or you are thinking about hurting yourself, help is available. Please call the Veterans Crisis Hotline at 988, send a text to 838255, or <u>click here</u> to access the Veterans Crisis Line.
- If questions in the study survey made you distressed or you want to talk to someone about how those questions

| | I consent/agree to participate |
|---|---|
| | clicking the button below, you are confirming that you have read all of the study information above and ree to participate in the study. |
| | ou may print this page for your records. You may also contact the study team to have a copy of this information ailed to you. |
| | PLEASE COMPLETE THE SURVEY ON A COMPUTER OR TABLET WITH INTERNET ACCESS, AS YOU MAY HAVE TROUBLE VIEWING THE SURVEY ON A MOBILE DEVICE. |
| • | If you aren't sure you are having an emergency and don't want to wait until regular business hours, you may also call the VA Boston HealthCare System at and ask the operator to page the psychiatrist on call. Tell the operator that you are a research participant. |
| • | If you need emergency care because you took part in this study, the VA will provide care to you. Be sure to tell the VA that you are in a research study. Please call 911 if you have a medical emergency. |
| • | If you want to talk to someone about your general rights as a study participant, please call the VA Boston Research Compliance Officer at |
| | made you feel, please call Dr. who is a clinical psychologist and a member of our research staff, at figure is unavailable, and you are in crisis, you are encouraged to go to your nearest emergency room. Otherwise, please leave a message, and she will return your call Monday-Friday within 24 hours. If you have a therapist, you might also want to discuss this study with him or her. |